CLINICAL TRIAL: NCT07152028
Title: Effects Of 6- Versus 12-Week Supervised Multimodal Exercise on Health Outcomes and Adherence in Obese Women: A Pilot Study
Brief Title: Exercise Supervision Duration and Adherence in Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Raziye Şavkın, Assoc.Prof., Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-60116787-020-237124
Record Dates: First submitted 2025-08-25; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Obesity (Disorder)
Keywords: obesity; exercise; Supervised exercise; Exercise adherence; Quality of life
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1= 6-week supervised plus 6-week home-based program (Other): Participants perform a 12-week multimodal exercise program targeting balance, muscular strength, core endurance, and cardiovascular fitness. Weeks 1-6 are supervised; weeks 7-12 are home-based via a video catalogue. Walking ≥30 min on ≥2 non-training days is encouraged.
  Interventions: Other: Exercise program with supervised and home-based components
- Group 2= Fully supervised 12-week program (Other): Participants perform a fully supervised 12-week multimodal exercise program including warm-up, balance, aerobic, strength, and core exercises. Walking ≥30 min on ≥2 non-training days is included.
  Interventions: Other: Fully supervised exercise program

INTERVENTIONS:
Other: Exercise program with supervised and home-based components — The 12-week program targets balance, muscular strength, core endurance, and cardiovascular fitness. Weeks 1-6 are supervised; weeks 7-12 are home-based via a video catalogue. Walking ≥30 min on ≥2 non-training days is advised. Intensity, repetitions, and sets are individualized using Borg CR-6-20. Adherence is monitored via exercise diaries and weekly phone calls with adjustments as needed.
  Arms: Group 1= 6-week supervised plus 6-week home-based program
Other: Fully supervised exercise program — The 12-week program is fully supervised and includes warm-up, balance, aerobic, strength, and core exercises. Walking ≥30 min on ≥2 non-training days is included. Intensity, repetitions, and sets are individualized using Borg CR-6-20. Adherence is monitored by a physiotherapist using exercise diaries.
  Arms: Group 2= Fully supervised 12-week program

SUMMARY:
Obesity is one of the most common health problems worldwide and is associated with many chronic diseases. Regular physical activity is known to play an important role in weight control, balance, quality of life, and mental health. However, obese individuals often have low adherence to exercise programs, and long-term maintenance of physical activity remains a major challenge.

Previous studies have shown that supervised exercise programs are effective in improving functional capacity and psychological well-being. On the other hand, home-based programs are less costly and more accessible, but adherence and effectiveness may be limited without professional supervision. To date, there is limited evidence on the optimal supervision duration needed to achieve sustainable improvements in obese women.

In the present study, it is aimed to investigate the effects of a 12-week individualized multimodal exercise program with different supervision durations (6 weeks supervised + 6 weeks home-based vs. 12 weeks fully supervised) on adherence and health outcomes in obese women. It is thought that prolonged supervision may increase exercise adherence, improve balance and functional performance, reduce depressive symptoms, and contribute positively to the quality of life. The results of this study may guide the design of future exercise programs for obesity management and provide evidence for more effective and sustainable rehabilitation approaches.

DETAILED DESCRIPTION:
Obesity is one of the leading public health problems worldwide and is strongly associated with cardiovascular diseases, diabetes, musculoskeletal disorders, and psychological problems. In addition to medical complications, obesity also negatively affects quality of life, daily activities, and mental well-being. According to epidemiological studies, the prevalence of obesity is steadily increasing, particularly among women, and this situation creates a serious burden on health systems.

Regular physical activity is one of the most effective non-pharmacological methods for the management of obesity. Exercise improves cardiovascular health, increases muscle strength, supports balance, reduces depressive symptoms, and contributes to weight control. Despite these benefits, adherence to exercise programs in obese individuals is often low, and sustaining physical activity over the long term remains a challenge.

Previous studies have reported that supervised exercise programs are more effective in ensuring adherence and providing functional and psychological benefits compared to unsupervised programs. However, home-based exercise programs are easier to access, more cost-effective, and provide flexibility in daily life. Nevertheless, lack of professional supervision may reduce motivation and exercise quality, leading to lower adherence and limited health benefits.

Physiotherapy and rehabilitation interventions for obesity generally include aerobic training, muscular endurance and strengthening exercises, posture and balance training, and core stabilization. Multimodal exercise programs that combine these approaches can improve both physical and psychological outcomes. Still, the optimal supervision duration in such exercise programs has not been clearly defined in the literature. While some studies emphasize the advantages of fully supervised training, others suggest that partial supervision combined with home-based practice may also be effective.

In this context, it is important to investigate whether extended supervision provides superior outcomes compared to a shorter period of supervision followed by home-based training. This information may help clinicians to design exercise programs that are both effective and sustainable for obese patients.

The present study aims to examine the effects of a 12-week individualized multimodal exercise program with different supervision durations (6 weeks supervised + 6 weeks home-based vs. 12 weeks fully supervised) in obese women. The investigators hypothesize that longer supervision will improve adherence, enhance functional capacity and balance, reduce depressive symptoms, and increase overall quality of life. The results of this study are expected to contribute to the development of more effective and practical rehabilitation approaches for the management of obesity.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years
* Body mass index (BMI) > 30 kg/m²

Exclusion Criteria:

* Clinically unstable cardiopulmonary disease (e.g., recent myocardial infarction, unstable angina)
* Musculoskeletal or neuromuscular disorders
* Cognitive impairments that could limit exercise participation
* Use of medications affecting bone metabolism

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Exercise adherence | 12 weeks
  Adherence to the exercise program was assessed by the percentage of completed exercise sessions recorded in exercise diaries (participant-reported), attendance checklists maintained by the supervising physiotherapist during supervised sessions, and weekly telephone follow-up logs during the home-based phase (weeks 7-12 for Group 1).

SECONDARY OUTCOMES:
Functional lower extremity strength | Baseline, 6 weeks, 12 weeks
  Assessed using the 30-second Chair Sit and Stand Test; higher repetitions indicate better functional strength.
Balance | Baseline, 6 weeks, 12 weeks
  Measured using the Timed Up and Go Test; shorter completion time indicates better balance and mobility.
Aerobic exercise capacity | Baseline, 6 weeks, 12 weeks
  Evaluated using the 6-minute Walk Test; longer walking distance indicates higher aerobic capacity.

OTHER OUTCOMES:
Health-related quality of life | Baseline, 6 weeks, 12 weeks
  Assessed using the Nottingham Health Profile (NHP); higher scores indicate poorer quality of life.
Depressive symptoms | Baseline, 6 weeks, 12 weeks
  Measured using the Beck Depression Inventory (BDI); higher scores indicate more severe depressive symptoms.
Physical activity level | Baseline, 6 weeks, 12 weeks
  Quantified using the International Physical Activity Questionnaire-Short Form (IPAQ-SF) in MET-min/week; higher scores indicate higher activity levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No